CLINICAL TRIAL: NCT05480514
Title: Clinical Evaluation of Daily Disposable Etafilcon A Cosmetic Contact Lenses
Brief Title: Clinical Evaluation of Daily Disposable Etafilcon A Cosmetic Contact Lenses (2022)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-6489
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Visual Acuity

STUDY DESIGN:
Masking Description: Brand masking: subjects, investigators, and clinical site personnel will be unaware of the identity (brand) of both study lenses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Eligible subjects will be randomized to the wear sequence (TEST/CONTROL) to wear the study lenses during each dispensing period (5 to 7 days) with a wash-out period (2 to 5 days) between wears.
  Interventions: Device: TEST LENS; Device: CONTROL LENS
- CONTROL/TEST (Experimental): Eligible subjects will be randomized to the wear sequence (CONTROL/TEST) to wear the study lenses during each dispensing period (5 to 7 days) with a wash-out period (2 to 5 days) between wears.
  Interventions: Device: TEST LENS; Device: CONTROL LENS

INTERVENTIONS:
Device: TEST LENS — etafilcon A with cosmetic pattern
Device: CONTROL LENS — Acuvue 1-Day Define Fresh Honey

SUMMARY:
This is a multi-site, 4-visit, brand-masked, bilateral, 2x2 cross-over dispensing study to evaluate visual acuity.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
2. Females between 18 and 29 (inclusive) years of age at the time of screening
3. Appear able and willing to adhere to the instructions set forth in this clinical protocol (i.e. willing to wear only the study lenses and not use habitual lenses during the dispensing periods)
4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last 30 days by self-report
5. Be a current wearer of cosmetic/circle lenses in the last 6 months, by self-report
6. The subject must be willing to be photographed and/or video-taped
7. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye
8. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye
9. Have spherical best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Currently pregnant or lactating
2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg, rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion)
3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion)
4. Any previous, or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.)
5. Any previous history or signs of a contact lens-related corneal inflammatory event (eg, past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear (at the investigators discretion).
6. Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment
7. Employee or family members of clinical site (eg, Investigator, Coordinator, Technician)
8. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion)
9. Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 89 (Actual)
Dates: Start 2022-08-27 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (2):
- Hong Kong (2):
  - Vital Eyecare Center Limited, Mong Kok, Kowloon
  - Sight Enhancement Center, Yau Ma Tei, Kowloon

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 89 subjects were enrolled in this study. Of those enrolled, 77 subjects were dispensed at least one study lens. Of those dispensed, 54 subjects completed the study while 23 subjects were discontinued.
Groups:
- Test [Etafilcon A] \ Control [Etafilcon A]: Subjects in this sequence were randomized to receive the Test [etafilcon A] lens during the first period and the Control [etafilcon A] lens during the second period.
- Control [Etafilcon A] \ Test [Etafilcon A]: Subjects in this sequence were randomized to receive the Control [etafilcon A] lens during the first period and the Test [etafilcon A] lens during the second period.
Period: Period 1
Arm/Group | Test [Etafilcon A] \ Control [Etafilcon A] | Control [Etafilcon A] \ Test [Etafilcon A]
Started | 38 | 39
Completed | 32 | 30
Not Completed | 6 | 9
Not completed — Pd-Incorrect Lens Power Assigned | 2 | 3
Not completed — Unsatisfactory Lens Fitting Due to Test Article | 3 | 5
Not completed — Subject No Longer Meets Eligibility Criteria | 0 | 1
Not completed — Covid-19 Related | 1 | 0
Period: Period 2
Arm/Group | Test [Etafilcon A] \ Control [Etafilcon A] | Control [Etafilcon A] \ Test [Etafilcon A]
Started | 32 | 30
Completed | 28 | 26
Not Completed | 4 | 4
Not completed — Unsatisfactory Lens Fitting Due to Test Article | 4 | 4

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects dispensed one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.4 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 77
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong, S.A.R., China | 77

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With LogMAR Visual Acuity Less Than 0.176 (20/30 Snellen Acuity)
Description: Visual acuity on logMAR (Logarithm of Minimal Angle of Resolution) scale was evaluated at distance (4 meters) under high luminance low contrast and low luminance high contrast lighting conditions using ETDRS (Early Treatment Diabetic Retinopathy Study) charts. Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. However, the data was dichotomized as Y=1 if logMAR visual acuity was less than 0.176 logMAR; and Y=0 otherwise. A value of 0.176 logMAR ≅20/30 Snellen Visual Acuity. The proportion of eyes with visual acuity lower than 0.176 logMAR was reported.
Time Frame: 5-minutes post-lens-fitting
Population: All subject dispensed at least one study lens.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Groups:
- Test [Etafilcon A]: Subjects that wore the Test [etafilcon A] lens during any of the two study periods.
- Control [Etafilcon A]: Subjects that wore the Control [etafilcon A] lens during any of the two study periods.
Arm/Group | Test [Etafilcon A] | Control [Etafilcon A]
Number analyzed (Participants) | 68 | 71
Number analyzed (Eyes) | 136 | 142
Proportion of eyes | 1 | 1
Statistical Analysis 1: Comparison: Test [Etafilcon A] vs Control [Etafilcon A]; Test type: Superiority — A superiority margin of 0.90 was used. Superiority was concluded if the lower bound of the 95% central posterior credible interval was above 0.90; Bayesian beta-binomial model; Mean Posterior Proportion = 0.9741, 95% CI 2-sided [0.9445 to 0.9926], Standard Deviation 0.01244

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; Approximately 3-weeks per subject
Groups:
- Test [Etafilcon A]: Subjects that wore the Test [etafilcon A] lens during any point in the study
- Control [Etafilcon A]: Subjects that wore the Control [etafilcon A] lens during any point in the study.
Arm/Group | Test [Etafilcon A] | Control [Etafilcon A]
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/71
Other Adverse Events (participants affected / at risk) | 0/68 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT05480514/Prot_SAP_000.pdf